CLINICAL TRIAL: NCT07055113
Title: Adapting Rehabilitation Delivery for Maximum Impact at Home-2 (ReDI-2)
Acronym: ReDI-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Pro00153489
Record Dates: First submitted 2025-06-20; First posted 2025-07-08 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Knee Osteoarthritis; Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: After providing consent, all participants will be assessed using standardized measures and then continue 12-weeks of community-based OA usual care. Following 12-weeks of usual care, they will be randomized to either of the intervention arms.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual Physical Therapy (IPT) (Experimental): 12-week virtual physical therapy that includes one-on-one visits with a physiotherapist.
  Interventions: Behavioral: Individual-based Virtual Physical Therapy Program
- Group-based Physical Therapy (GPT) (Experimental): 12-week virtual physical therapy that includes group classes (4-5 participants) with two physiotherapists. In each session, each participant will also have a 10-12 min one-on-one interaction with one of the physiotherapists.
  Interventions: Behavioral: Group-based Virtual Physical Therapy Program

INTERVENTIONS:
Behavioral: Individual-based Virtual Physical Therapy Program — Twelve-week virtual physical therapy that includes one-on-one visits with a physiotherapist.
  Multi-modal Self-management program comprises:
  * Education to understand OA and its management: 'Understanding & Managing OA'; 'Activity & Exercise'; 'Managing Pain'; 'Healthy Eating'; 'Mental & Emotional Well-being'; 'General Wellness'.
  * Personalized Goal Setting in partnership with therapist to promote patient activation.
  * Progressive neuro-muscular exercises of the core and lower extremity, customized to patient capacity with participants encouraged to perform exercises at least 2 times/week between PT sessions to improve strength and function; 2 levels of resistance bands will be provided to progress resistance.
  * Physical activity goals using FitBit step count, to increase daily activity as tolerated.
  Arms: Individual Physical Therapy (IPT)
Behavioral: Group-based Virtual Physical Therapy Program — Twelve-week virtual physical therapy that includes group classes (4-5 participants) with two physiotherapists. In each session, each participant will also have a 10-12 min one-on-one interaction with one of the physiotherapists.
  Multi-modal Self-management program comprises:
  Education to understand OA and its management: 'Understanding & Managing OA'; 'Activity & Exercise'; 'Managing Pain'; 'Healthy Eating'; 'Mental & Emotional Well-being'; 'General Wellness'.
  Personalized Goal Setting in partnership with therapist to promote patient activation.
  Progressive neuro-muscular exercises of the core and lower extremity, customized to patient capacity with participants encouraged to perform exercises at least 2 times/week between PT sessions to improve strength and function; 2 levels of resistance bands will be provided to progress resistance.
  Physical activity goals using FitBit step count, to increase daily activity as tolerated.
  Arms: Group-based Physical Therapy (GPT)

SUMMARY:
People who live in rural areas and have hip or knee arthritis can have difficulty receiving physical therapy (PT) close to home. Living with hip or knee arthritis can make doing daily activities and being physically active difficult. This can lead to other health conditions, such as becoming overweight, or lessen enjoyment of life.

We will compare 2 programs that allow physical therapists to treat rural residents in their own home to each other and to usual care. Usual care is the care that is typically provided to people living with hip or knee arthritis.

For the first 12 weeks, participants will continue usual osteoarthritis (OA) care and then complete the standardized questionnaires again. Then, they will be randomized to either Individual (IPT) or Group-based PT (GPT).

Over 12-weeks, therapists will meet virtually with patients using Zoom so that patients and therapists can see each other. The program will be either a class or one-on-one with a therapist. In the class, participants will still receive private one-to-one time with the therapist using a Zoom 'breakout' room. Therapists in both groups will help patients do exercises correctly in their home. Patients can also see and talk to the therapists to discuss their challenges in living with OA and set personalized goals including pain management, participating in valued daily activities, keeping healthy (diet, sleep) and being active. Both programs will allow patients who sometimes cannot access physical therapy to receive care in their home.

DETAILED DESCRIPTION:
Adapting Rehabilitation Delivery for Maximum Impact at Home-2 (ReDI-2) is a randomized clinical trial (RCT) that will assess the impact of 12-weeks of community-based osteoarthritis (OA) usual care and then compare two 12-week virtual home-based rehabilitation programs (IPT or GPT) for rural Albertans living with hip and/or knee OA to each other and to usual care. ReDI-2 aims to improve self-management through patient activation. Program content will be identical with only the delivery format differing between groups.

IPT will be one-to-one virtual PT for OA self-management including education, exercise and personalized goal-setting, including physical activity goals.

GPT will use 2 PTs and 4-5 participants/class. One therapist will provide personalized goal-setting with each participant via a Zoom 'breakout' room, while the 2nd therapist leads group-based therapy in the 'main' Zoom room comprised of education and exercises individualized to participants' capacity.

Objectives and Hypotheses Primary Objective: To compare the effectiveness of 12-weeks of virtual IPT or GPT, to each other and to 12-weeks of usual care, in rural Albertans living with hip or knee OA, on changes in self-management measured through patient activation, using the validated 13-item Patient Activation Measure (PAM).

Secondary Objectives: 1) To compare the effectiveness of a) virtual IPT and GPT to each other and to usual care post-intervention in rural Albertans living with hip or knee OA in terms of HRQL, understanding pain management, improving step count (as a measure of physical activity), pain, and function, including physical performance, and b) primary and secondary outcomes up to 12-months post-intervention; and 2) To explore how patient and program characteristics affect outcomes in each model, which may highlight responders/non-responders.

Research Method/Procedures Design. ReDI-2 is a randomized parallel-arm, single-blind (clinical assessor) trial.

OA Usual Care. After providing consent, all participants will be assessed using standardized measures and then continue 12-weeks of community-based OA usual care, including the screening clinics' educational materials that encourage exercise, physical activity and wellness, and any community-based treatments that patients independently seek (uncommon). Investigators are not including a usual care only group due to low impact and reported attrition rates of about 25%, so investigators will evaluate all participants at trial entry and 12-weeks later to observe the impact of usual care. Usual care is the same duration as the ReDI-2 interventions so that investigators do not under-estimate potential benefits of usual care.

Virtual Home-Based Interventions. Following 12-weeks of usual care, the research coordinator will randomize participants to IPT or GPT. A technology support person will call participants to set up Zoom and prepare for PT sessions. Participants not using a laptop will attach their cellphone or tablet to a provided selfie-stick. Participants will receive an email with an embedded link to connect to a secure Zoom session that connects their camera, microphone and speaker to the provider's device.

Our multi-modal Self-management program comprises:

Education to understand OA and its management: Week 1 (W1) 'Understanding & Managing OA'; (W2) 'Activity & Exercise' (when participants are afraid to move, exercising when participants have pain & OA); (W3) 'Managing Pain' (medications including inappropriateness of opioid use, heat/ice, pacing & conserving energy, bracing & mobility aides to promote activity); (W4) 'Healthy Eating' (weight & OA, know the portions, nutrition for bone health); (W5) 'Mental & Emotional Well-being' (managing stress, depression, & anxiety); (W6) 'General Wellness' (sleep, dental health, quitting smoking). Educational materials will be offered in paper and e-formats.

Personalized Goal Setting in partnership with their therapist using Specific, Measureable, Attainable, Relevant, Time-based (SMART) goals to promote patient activation.

Progressive neuro-muscular exercises of the core and lower extremity, customized to patient capacity with participants encouraged to perform exercises at least 2 times/week between PT sessions to improve strength and function; 2 levels of resistance bands will be provided to progress resistance. Physical activity goals using FitBit step count, to increase daily activity as tolerated.

Program Frequency and Duration: Both IPT and GPT groups will have weekly sessions for 6 weeks, followed by a 2-week break to encourage participants to manage their OA independently, and promote retention of new behaviours. Participants will then return at 9 weeks to progress exercises and goals. A second optional 'check-in' visit at 12 weeks will assess uptake of participants' expressed desire to have more check-ins with therapists as they gain confidence in self-management.

IPT sessions will each be about 45 minutes; therapists will discuss OA self-management, review and advance SMART goals, progress exercises and encourage exercise performance between sessions and set step count goals.

GPT sessions will each last about 75-90 minutes. All participants (4 to 5/session) will initially join the 'main' Zoom room to receive educational content from both therapists and encourage participant networking (about 10-15 minutes). One therapist will then move to the 'breakout' room, with each participant joining the 'breakout room' for 10-12 minutes of one-to-one SMART goal-setting, and review and progression of physical activity goals. Therapists will coordinate transitions between the 'main' room and the 'breakout' room. To develop a therapeutic relationship with each participant, the same therapist will lead all breakout sessions. In the 'main' room, the 'Exercise' therapist will use a 36-inch monitor to visualize all participants to correct and progress exercise performance. In the final 5 minutes, all participants and both therapists will join the 'main' room to review the session; participants will be encouraged to perform exercises twice between group sessions.

Recruitment. The Edmonton Bone and Joint (Edmonton) Clinic will serve as our recruitment centre as they see high volumes of potentially eligible patients, who, when deemed non-surgical, are often seeking treatment resources.

Screening: Clinic staff will identify eligible patients (OA diagnosis and rural address) and determine their interest in the study. Research personnel will confirm eligibility and obtain signed consent.

Selection Criteria: Eligible patients will: have confirmed hip or knee OA, but deemed to not require TJR (i.e., not on the surgical waitlist); not currently be attending PT; reside outside of Edmonton or nearby communities; be English-speaking with access to a Zoom-friendly device (smart phone, tablet, laptop). Those reporting uncontrolled co-morbidities (e.g., hypertension, diabetes) will seek clearance to participate from their family physician.

Enrollment: Following consent, all participants will receive information provided by the screening clinics as per usual care regarding OA management. Approximately 10 weeks after enrollment, the technology support person will call participants to install Zoom on their selected device and provide instructions, and then mail out the remaining study items as needed, at no cost to participants (tripod selfie-stick to hold their smart phone or tablet, FitBit, and 2 resistance bands of varying intensity).

Research evaluations will be undertaken by the blinded assessor, will occur at pre-usual care, pre-intervention (post-usual care), immediate post-intervention, and 6- and 12-months post-intervention. Participants will be encouraged to wear the FitBit daily both during and after the intervention, but instructed to wear it for 14 weeks (i.e., one-week before and after, as well as during the intervention period) and then for at least 1 week before research assessments to measure step count using the FitBit Dashboard. As a FitBit is not OA usual care, investigators will be unable to assess step count during usual care as providing a FitBit could act as an intervention, artificially inflating step count during the usual care period, even without coaching.

ELIGIBILITY:
Inclusion Criteria:

* Patient with confirmed hip or knee OA, but deemed to not require total joint arthroplasty (i.e., not on the surgical waitlist)
* Not currently be attending physiotherapy
* Reside outside of Edmonton or nearby communities
* English-speaking
* with access to a Zoom-friendly device (smart phone, tablet, laptop).

Exclusion Criteria:

• Patients who are not meeting the inclusion criteria are not eligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Activation Measure (PAM) | pre-usual care, pre-intervention, immediate post-intervention, 6-months post-intervention,12-months post-intervention
  Self-management will be measured using the validated 13-item Patient Activation Measure (PAM). Responses are scored to a total score on a 0-100-point scale with higher scores representing higher patient activation.

SECONDARY OUTCOMES:
Pain - Numeric Rating Scale (NRS) | pre-usual care, pre-intervention, immediate post-intervention, 6-months post-intervention,12-months post-intervention
  Pain will be assessed using the Numeric Rating Scale. Responses are scored to a total score on a 0-10 point scale with higher scores representing more pain.
Pain Catastrophizing Scale (PCS) | pre-usual care, pre-intervention, immediate post-intervention, 6-months post-intervention,12-months post-intervention
  Negative cognitive & emotional responses to actual or anticipated pain will be assessed via the Pain Catastrophizing Scale. Responses are scored to a total score of 0-52 with a higher score reflecting more catastrophizing thoughts.
Knee Osteoarthritis Outcome Score (KOOS) - Health-Related Quality of life (HRQL) | pre-usual care, pre-intervention, immediate post-intervention, 6-months post-intervention,12-months post-intervention
  Health-related quality of life (HRQL) will be assessed via the validated Knee Osteoarthritis Outcome Score (KOOS). Responses are summed on a 0-100-point scale, with lower score representing worse problems.
Knee Osteoarthritis Outcome Score (KOOS) - Daily Living Function | pre-usual care, pre-intervention, immediate post-intervention, 6-months post-intervention,12-months post-intervention
  Daily Living Function will be assessed via the validated Knee Osteoarthritis Outcome Score (KOOS). Responses are summed on a 0-100-point scale, with lower score representing worse problems.
Hip Osteoarthritis Outcome Score (HOOS) - Health-Related Quality of life (HRQL) | pre-usual care, pre-intervention, immediate post-intervention, 6-months post-intervention,12-months post-intervention
  Health-related quality of life (HRQL) will be assessed via the validated Hip Osteoarthritis Outcome Score (HOOS). Responses are summed on a 0-100-point scale, with lower score representing worse problems.
Hip Osteoarthritis Outcome Score (HOOS) - Daily Living Function | pre-usual care, pre-intervention, immediate post-intervention, 6-months post-intervention,12-months post-intervention
  Daily Living Function will be assessed via the validated Hip Osteoarthritis Outcome Score (HOOS). Responses are summed on a 0-100-point scale, with lower score representing worse problems.
Euro-Quality of Life-5 Dimension-5 Level (EQ-5D-5L) | pre-usual care, pre-intervention, immediate post-intervention, 6-months post-intervention,12-months post-intervention
  Health status will be assessed using the validated EuroQoL-5 Dimension-5 Level (EQ-5D-5L). It consists of 2 parts: 1.EQ-5D-5L: self-report, generic health utility instrument with 5 domains (mobility, self-care, pain/discomfort, depression/anxiety, and usual activities) and 5 levels in each domain (no problems, slight problems, moderate problems, severe problems, and extreme problems). 2. EQ Visual Analogue scale (EQ VAS): Scores: 100 = the best health you can imagine and 0 = the worst health you can imagine.
30-second Chair Stand test | pre-intervention, immediate post-intervention, 6-months post-intervention,12-months post-intervention
  Lower extremity strength / balance will be measured using the 30-second Chair Stand test modified and validated for virtual use. The number of sit-to-stands that participant completes in 30 seconds is recorded.
Fitbit Step count | pre-intervention, immediate post-intervention, 6-months post-intervention,12-months post-intervention
  Physical activity will be assessed using Fitbit step count. The avearge number of steps per day will be recorded.
Global rating of change/pain - Patient | pre-intervention (post-usual care), immediate post-intervention, 6-months post-intervention,12-months post-intervention
  Patient's ability to self-manage pain will be assessed via the Global rating of change/pain. It is scored on a 7- point scale (1 Much better - 7 Much worse).
Global rating of change/function - Patient | pre-intervention (post-usual care), immediate post-intervention, 6-months post-intervention,12-months post-intervention
  Patient's ability to function will be assessed via the Global rating of change/function. It is scored on a 7- point scale (1 Much better - 7 Much worse).
Global rating of change/physical activity - Patient | pre-intervention (post-usual care), immediate post-intervention, 6-months post-intervention,12-months post-intervention
  Patient's ability to be physically active will be assessed via the Global rating of change/physical activity. It is scored on a 7- point scale (1 Much better - 7 Much worse).
Global rating of change/OA self-management - Patient | pre-intervention (post-usual care), immediate post-intervention, 6-months post-intervention,12-months post-intervention
  Patient's ability to self-manage arthritis will be assessed via the Global rating of change/OA self-management. It is scored on a 7- point scale (1 Much better - 7 Much worse).
Global rating of change/satisfaction - Patient | pre-intervention (post-usual care), immediate post-intervention, 6-months post-intervention,12-months post-intervention
  Patient's satisfaction will be assessed via the Global rating of change/satisfaction. It is scored on a 7- point scale (1 Very satisfied - 7 Very dissatisfied).
Telehealth Usability Questionnaire - Patient | immediate post-intervention
  Patient experience will be assessed via the validated Telehealth Usability Questionnaire. The responses are scored on a 5- point scale (1 Strongly disagree - 5 Strongly agree).
Global rating of change/satisfaction - Provider | immediate post-intervention
  Provider's satisfaction will be assessed via the Global rating of change/satisfaction. It is scored on a 7- point scale (1 Very satisfied - 7 Very dissatisfied).
Telehealth Usability Questionnaire - Provider | immediate post-intervention
  Provider experience will be assessed via the validated Telehealth Usability Questionnaire. The responses are scored on a 5- point scale (1 Strongly disagree - 5 Strongly agree).

CONTACTS AND LOCATIONS:
Locations (1):
- Edmonton Bone and Joint Centre, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
We are working with our ethics board to determine what level of deidentified data we can release based on criteria such as the size of our analytic cells.